CLINICAL TRIAL: NCT05046444
Title: Testing the Diagnostic Supremacy of Sequencing-only Approaches in Hematologic Malignancies: an Observational Trial
Brief Title: Solving Riddles Through Sequencing
Acronym: SIRIUS
Status: Recruiting | Type: Observational
Sponsor: Munich Leukemia Laboratory (Industry)
Collaborators: Illumina, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MLL_002
Record Dates: First submitted 2021-07-22; First posted 2021-09-16 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Leukemia; Hematologic Malignancy; Rare Diseases; Refractory Leukemia; Refractory Lymphoma; Unknown Primary Tumors
MeSH Terms: conditions — Leukemia; Hematologic Neoplasms; Rare Diseases; Lymphoma; Neoplasms, Unknown Primary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood smears for morphology and/or peripheral blood or bone marrow for immunophenotyping from all hematological malignancies recognized by current WHO classification (Swerdlow et al. 2017)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unclear diagnosis via conventional methods: The study population consists of carefully chosen patients with potential hematological malignancy, for which current diagnostic methods were not sufficient to provide clear-cut diagnosis and definitive clinical guidance. SIRIUS will be conducted for a total number of 110 patients with inconclusive diagnosis by gold standard techniques for a total of up to nine months after the first enrollment.
  Interventions: Diagnostic Test: Next Generation Sequencing

INTERVENTIONS:
Diagnostic Test: Next Generation Sequencing — NON-Interventional Observation only study comparing sequencing-only approaches to classical diagnostic methods
  Other Names: NGS, Whole genome Sequencing

SUMMARY:
During the last decades hematologists have excelled at improving and refining the classification, diagnosis, and thus ultimately the therapeutic decision-making process for their patients. This continuous evolution proceeded in parallel to seminal discoveries in basic science such as FISH, PCR and NGS. So far, the current WHO classification serves as reference to diagnostic decision making and is largely based on 5 diagnostic pillars: cytomorphology of peripheral blood and/or bone marrow smears, histology and immunohistochemistry of bone marrow trephine biopsies or lymph nodes, immunophenotyping, chromosome banding analysis supplemented by FISH analysis, molecular genetics including PCR and targeted panel sequencing via NGS. This leads to a swift diagnosis in 90 % of all cases. The leftover 10 % remain a challenge for hematopathologists and clinicians alike and are resolved through interdisciplinary teams in the context of specialized boards. With the advent of high throughput sequencing (mainly WGS and WTS) the possibility of a comprehensive and detailed portrait of the genetic alterations - specifically in challenging cases - has become a realistic alternative to classical methods. In SIRIUS the investigators will prospectively challenge this hypothesis to address the question of how often a better or final diagnosis can be delivered by WGS and/or WTS and if unclear cases can be efficiently resolved.

DETAILED DESCRIPTION:
1. Background and Rationale Treatment of hematological diseases relies on a single cardinal prerequisite: correct classification within the broad specter of malignant diseases arising from the hematopoietic system. With the ever-expanding availability of distinct yet complementary diagnostic tools, our understanding of the landscape of hematological diseases steadily increases. As such, the current consensus classification as summarized through the WHO classification (2017) represents a compass guiding diagnostic algorithms to the correct diagnosis. Today, the gold standard of routine diagnostic process relies on five methodological pillars: cytomorphology, histology, chromosomal cytogenetics, immunophenotyping, and molecular genetic testing. This leads to a treatment enabling diagnosis in the vast majority of cases. However, approximately 10 % of cases remain unresolved from a diagnostic point of view and hence do not lead to a satisfactory diagnosis according to current WHO standards (2017). The investigators intend to solve this issue to provide illuminating diagnostic guidance for the best possible patient´s care.
2. Objectives To address this problem, the investigators hypothesize that novel high throughput sequencing methods, e.g., whole genome and/or whole transcriptome sequencing are able - by virtue of painting a more delicate genetic portrait of a tumor sample - to provide a more accurate diagnosis.

To this end the investigators generated a reference collection of 5,500 samples with the full spectrum of hematological malignancies, for which the investigators performed whole-genome sequencing as well as whole-transcriptome sequencing. Moreover, gold standard diagnoses according to WHO classification with all needed techniques, all performed in MLL, clinical data and therapy response data are fully available for these cases. The main advantage of this reference collection consists of the unambiguity of each diagnosis, providing a reference framework for any further classification and diagnosis especially in difficult cases.

Therefore, SIRIUS will compare the diagnostic superiority of WGS or WTS to the combined approach with gold standard results and by matching the obtained results to the nearest "digital sibling" within our reference cohort of more than 5,500 WGS and WTS (both in 93% of cases). To this end, the investigators will use an inhouse developed matching algorithm, which is able to match genomic or transcriptomic profiles to a group of similar cases and gold standard results from timepoint of this study. Current workflows intended to generate WTS/WGS data from patient samples - all while fulfilling state of the art accreditation (ISO 15189) - require up to 5 - 7 days. This is largely comparable to classical methods but holds the promise to replace error prone and arduous iterations in the methodological work up. The objective is to test whether WTS and/or WGS based approaches can surpass classical methods regarding diagnostic precision and routine reliability. Here the investigators will test this hypothesis in a prospective real-world setting under diagnostically difficult circumstances.

ELIGIBILITY:
Inclusion Criteria:

* Patients having been investigated with a suspected hematological disorder and:
* Having unclear diagnosis after internal routine diagnosis
* Unusual clinical course
* Unusual r/r status or non-responder
* Multiple parallel hematological conditions
* Difficult/rare therapy associated/secondary neoplasms
* Current diagnostic workup is not satisfactory in terms of (1) accuracy (2) clinical behavior
* Only samples of patients min. 18 years of age will be used
* Material with a minimum of 20% tumor content in bone marrow or peripheral blood sample
* Patient´s informed consent

Exclusion Criteria:

* Sample is not fit for state-of-the-art diagnosis, fails initial quality control. For quality insurance we will exclude samples with wrong anticoagulant sent. Samples with damage due to meteorological reasons (freeze-thaw damage or elevated temperature) will be excluded.
* Samples with to scarce material jeopardizing routine gold-standard diagnosis will be excluded (tumor content < 20 %).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SIRIUS is conducted as a monocentric prospective case-control study. The study population consists of carefully chosen patients with potential hematological malignancy, for which current diagnostic methods were not sufficient to provide clear-cut diagnosis and definitive clinical guidance. SIRIUS is entirely a non-interventional study without therapeutic consequences for direct patient care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
sequencing only versus gold standard diagnosis | Time Frame of Outcome: At diagnosis for each case/patient throughout the complete duration of study for approximately 1 year.
  The primary endpoint will be assessed as follows: unclear cases will be subjected to three diagnostic algorithms:
  1. Inhouse at referring site by histopathological diagnosis in the context of a hematological tumor board according to current standards
  2. Current gold-standard diagnostic workup as performed routinely by the MLL
  3. WGS and WTS sequencing plus matching to nearest digital sibling in 5,5k cohort
  We will compare the accuracy for approach #3 for each patient/case by comparing the sequencing results with the therapy guiding approach in domo and Current gold-standard diagnostic workup as performed routinely by the MLL. Accuracy and overlap or discordance will be measured in percentage (%) of total cohort. Time Frame of Outcome: At diagnosis for each case/patient throughout the complete duration of study for approximately 1 year.

SECONDARY OUTCOMES:
turnaround time | The time frame will be consisting of an assessment at diagnosis for next 14 days per case/patient.
  Turnaround time until potential therapy guiding diagnosis will be measure and compared in days.
actionable targets | This outcome will be measured one year after diagnosis. (1 year after diagnosis)
  The number of potential actionable targets will be determined for each case. We will assess this number in absolute numbers for each patient and for which a therapy has been approved but identification was missed in during classical gold standard diagnosis.
disease stage | This outcome will be measured one year after diagnosis. (1 year after diagnosis)
  We will Identify the putative disease stage based on sequencing only approaches in comparison to normal gold standard diagnosis as well as clinical history. Results will be denoted as percentage (%) of correctly classified cases.
Micro-cost analysis | The estimated timeframe for this outcome will be the timepoint of diagnosis for each patient (approximately 5 days)
  We will measure all costs for respective assays and personnel to finally compare workflows 2 and 3 (see primary outcome 1.).

CONTACTS AND LOCATIONS:
Locations (1):
- MLL Munich Leukemia Laboratory, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT05046444/Prot_000.pdf